CLINICAL TRIAL: NCT03801434
Title: Phase 2 Study of Ruxolitinib in Idiopathic Hypereosinophilic Syndrome and Primary Eosinophilic Disorders
Brief Title: Ruxolitinib in Treating Patients With Hypereosinophilic Syndrome or Primary Eosinophilic Disorders
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: William Shomali (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor-Investigator, William Shomali, Clinical Assistant Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-47457; NCI-2018-03723 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HEMMPD0035 (Other: Stanford Cancer Institute Palo Alto); IRB-47457 (Other: Stanford IRB)
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: BCR-JAK2 Fusion Protein Expression; Blasts 20 Percent or Less of Peripheral Blood White Cells; Blasts More Than 5 Percent of Bone Marrow Nucleated Cells; Blasts More Than 5 Percent of Peripheral Blood White Cells; Blasts Under 20 Percent of Bone Marrow Nucleated Cells; Chronic Eosinophilic Leukemia, Not Otherwise Specified; Eosinophilia; Hepatomegaly; Hypereosinophilic Syndrome; JAK2 Gene Mutation; Splenomegaly; TEL-JAK2 Fusion Protein Expression
MeSH Terms: conditions — Hypereosinophilic Syndrome; Eosinophilia; Hepatomegaly; Splenomegaly | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ruxolitinib) (Experimental): Patients receive ruxolitinib PO BID on days 1-28. Treatment repeats for up to 6 cycles (28 days each) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Given PO
  Other Names: INCB-18424; INCB18424; Oral JAK Inhibitor INCB18424

SUMMARY:
This phase II trial studies how well ruxolitinib works in treating patients with hypereosinophilic syndrome or primary eosinophilic disorders.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall hematologic response rate to ruxolitinib in patients with hypereosinophilic syndrome and primary eosinophilic disorders.

SECONDARY OBJECTIVES:

I. To determine safety profile of ruxolitinib in patients with hypereosinophilic syndrome and primary eosinophilic disorders.

II. To determine the proportion of patients on corticosteroids who are able to become corticosteroid-independent and/or reduce the dose by >= 50%.

III. To evaluate the duration of response (DoR). IV. To evaluate the time-to-response (TTR). V. To evaluate progression-free survival (PFS) and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Subject with idiopathic hypereosinophilic syndrome must meet the following:

  * Has as at least 2 readings with an absolute eosinophil count >= 1,500/mm^3 in the preceding 3 months prior to starting ruxolitinib (one reading must be during the screening period).
  * Dependent, intolerant or refractory to corticosteroids OR has relapsed/refractory disease to other therapy besides corticosteroids.
  * Symptomatic from his/her disease OR has one or more signs of organ damage (assessed by the investigator as possibly-related to eosinophilia or biopsy-proven). This can include skin, lung, cardiac, central nervous system, liver, or gastrointestinal (GI) involvement, or evidence of symptomatic hepatic or splenic enlargement.
* Subject with lymphocyte-variant hypereosinophilia must meet the following

  * Has at least 2 readings with an absolute eosinophil count >= 1,500/mm^3 in the preceding 3 months prior to starting ruxolitinib (one reading must be during the screening period).
  * Dependent, intolerant or refractory to corticosteroids* OR has relapsed/refractory disease to other therapy besides corticosteroids.
  * Symptomatic from his/her disease OR has one or more signs of organ damage (assessed by the investigator as possibly-related to eosinophilia or biopsy-proven). This can include skin, lung, cardiac, central nervous system, liver, or GI involvement, or evidence of symptomatic hepatic or splenic enlargement
  * Has abnormal T-lymphocyte immuno-phenotype by flow cytometry.
* Subject with chronic eosinophilic leukemia, not otherwise specified (CEL,NOS) must meet the following

  * Has at least 2 readings with an absolute eosinophil count >= 500/mm^3 in the preceding 3 months prior to starting ruxolitinib (one reading must be during the screening period).
  * Newly-diagnosed OR receiving corticosteroids OR has relapsed/refractory disease to any therapy besides corticosteroids.
  * Has increased blasts in the blood or bone marrow (> 5% and < 20%), and/or a clonal cytogenetic or molecular abnormality

    * Subjects with JAK2 mutations are included within this group.
* Subject with JAK2-rearranged eosinophilic neoplasm must meet the following

  * Has at least 2 readings with an absolute eosinophil count >= 500/mm^3 in the preceding 3 months prior to starting ruxolitinib (one reading must be during the screening period).
  * Newly-diagnosed OR receiving corticosteroids OR has relapsed/refractory disease to any therapy besides corticosteroids.

    * This group includes subjects with PCM1-JAK2, BCR-JAK2, ETV6-JAK2 or other JAK2 rearrangements.
* If receiving corticosteroids, must be a stable dose for >= 28 days prior to Day 1 (unstable dosing not eligible).
* Eastern Cooperative Oncology Group (ECOG) performance status =< 3.
* Willing and able to review and execute informed consent (legally-authorized consent acceptable).

Exclusion Criteria:

* Active life-threatening complication(s) from underlying eosinophilic disease (i.e., leukostasis; acute thromboembolic disease including central nervous system (CNS) involvement; severe pulmonary or cardiac dysfunction). Stabilization of acute, life-threatening eosinophil-related co-morbidities will allow enrollment of the patient.
* World Health Organization (WHO)-defined myeloid neoplasm associated with eosinophilia other than CEL NOS and JAK2 rearranged neoplasms (e.g., myelodysplastic syndrome (MDS); myeloproliferative neoplasms (MPN); MDS/MPN overlap disorders; and systemic mastocytosis (SM).
* Reactive hypereosinophilia due to connective tissue disease, sarcoidosis or eosinophilic granulomatosis with polyangiitis.
* Organ-restricted ?tissue? eosinophilia with the absence of peripheral eosinophilia in the blood.
* Invasive malignancy over the previous 2 years except treated early stage carcinomas of the skin, completely resected intraepithelial carcinoma of the cervix, and completely resected papillary thyroid and follicular thyroid cancers.
* Myeloid or lymphoid neoplasm with eosinophilia and abnormalities of PDGFRA, PDGFRB or FGFR1.
* Anticipated to receive a hematopoietic stem cell transplant within the first 6 months of treatment on trial.
* Major surgery within 4 weeks prior to entering the study.
* Life expectancy of < 6 months.
* Known diagnosis of human immunodeficiency virus (HIV).
* Known diagnosis of chronic active hepatitis B or C (viral testing is not required). Subjects with a known history of hepatitis B and/or C are allowed on trial if at the time of enrollment, the virus is not active and undetected (testing required if there is a known history), and such patients are not actively receiving antiviral treatment specific for hepatitis B and/or C.
* Clinically serious infections requiring ongoing antibiotic therapy.
* Parasitic infection diagnosed within 24 weeks prior to enrollment.
* Platelet count =< 25 x 10^9/L at baseline.
* Alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) > 4 x upper limit of normal (ULN) or direct bilirubin > 4 x ULN (if considered to be unrelated to the underlying eosinophilic disorder).
* End-stage renal function (creatinine clearance [CrCl] < 15 mL/min or glomerular filtration rate [GFR] < 15 mL/min) regardless of whether hemodialysis is required.
* Use of investigational or commercial therapies with the intent to treat the underlying eosinophilic disorder within 28 days of study start, including interferon; imatinib; alemtuzumab; cyclosporine; methotrexate; mepolizumab; benralizumab; or other antibody therapies.
* Use of hydroxyurea within 7 days of study start.
* Prior therapy with ruxolitinib or other JAK inhibitors.
* Previous allergic reactions to JAK inhibitors or excipients.
* Unwilling to commit to abstinence from heterosexual contact or agree to use and comply with highly effective contraception, 28 days prior to starting study drug, during the treatment period and for 12 weeks after discontinuation of study treatment.
* Females of childbearing potential who have a positive pregnancy test (urine or serum) during screening period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 3 years
  ORR is the sum of complete response (CR) plus complete response with incomplete platelet recovery (CRp) plus partial response (PR). Complete response, with platelet incomplete platelet recovery (CRp) is defined as a response that meets CR criteria but platelet count remains below 100 x 10^9/L. This outcome will be reported as a number.
  * Complete response (CR) = normalization of white blood cell (WBC) count; absolute eosinophil count in blood; and % eosinophils in blood, without increased blasts or eosinophils in bone marrow, and with a non-palpable spleen and/ or normal spleen size by imaging.
  * Partial response (PR) is defined as ≥ 50% reduction (if above normal range) in all the following: total WBC count; absolute eosinophil count in blood; % eosinophils in blood; % eosinophils and myeloblasts in bone marrow; in addition to spleen size reduction of ≥ 50% by palpation and/ or ≥35% by imaging (if increased at baseline).

SECONDARY OUTCOMES:
Adverse events | 3 years
  Adverse events will be reported including severity, seriousness, and relatedness of adverse events based on National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The outcome will be reported as a number of all serious adverse events; with frequency ≥ 10%.
Proportion of subjects who become corticosteroid-independent | 3 years
  Descriptive analysis of the proportion of subjects who become corticosteroid-independent for 12 or more consecutive weeks will be reported. The outcomes will be reported as number
Proportion of patients who reduce corticosteroid dose by >= 50% (including patients who become corticosteroid-independent) | 3 years
  Descriptive analysis of the proportion of subjects who reduce corticosteroid dose by >= 50% (including patients who become corticosteroid-independent) for 12 or more consecutive weeks will be reported. The outcomes will be reported as number
Duration of response (DoR) | 3 years
  Median duration of response (DoR) defined as the time from first onset of confirmed response to the date of first documented and confirmed progression or death due to hypereosinophilic syndrome or a primary eosinophilic neoplasm. This outcome will be reported as the median with full range, for those subjects that achieve a clinical response. Response defined as per the Primary Outcome.
Time to response (TTR) | 3 years
  Median time to response (TTR) is defined as the time from start of treatment until the date of onset of a confirmed response. This outcome will be reported as the median with full range, for those subjects that achieve a clinical response.
Median Progression-free survival (PFS) | 3 years
  Median progression free survival (PFS) is defined as the time from start of treatment to the date of the first documented and confirmed progression or death or institution of new therapy. This outcome will be reported as the median with full range. Progression is defined as ≥ 25% in one of the following when compared to baseline: total WBC count; absolute eosinophil count in blood; or % eosinophils in blood; OR the presence of ≥ 20% blasts in the peripheral blood or bone marrow ("evolution to AML"), with any lab finding confirmed at 2 weeks; or ≥ 25% increase in spleen size.

CONTACTS AND LOCATIONS:
Overall Officials: William E Shomali, MD, Principal Investigator — Stanford Cancer Institute Palo Alto
Locations (4):
- United States (4):
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - OHSU Knight Cancer Institute, Portland, Oregon
  - University of Utah, Salt Lake City, Utah
  - Fred Hutchinson cancer research center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No